CLINICAL TRIAL: NCT03343925
Title: Direct-acting Antiviral Therapy and Reinfection Among People With Chronic Hepatitis C Virus Infection and Recent Injecting Drug Use in Community-based Settings: the SHARP-C Study
Brief Title: Direct-acting Antiviral Therapy and Reinfection Among PWID With Chronic HCV in Community-based Settings
Acronym: SHARP-C
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP1605
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Reinfection
MeSH Terms: conditions — Hepatitis C, Chronic; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Plasma, PBMCs, Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SHARP-C is an observational cohort study investigating the effect of direct-acting antiviral (DAA) therapy and reinfection in people with chronic hepatitis C virus (HCV) and recent injecting drug use. A prospective, observational cohort design will be used to enrol patients attending tertiary drug and alcohol and primary health care services.

Participants will be prescribed a direct-acting HCV medication as per the standard of care. The on treatment phase will vary dependent on the type of a direct-acting antiviral prescribed as per the standard of care. Once patients have completed their treatment course they will be followed up every 3 months for up to 3 years following the end of treatment phase.

The study will aim to evaluate the incidence of HCV reinfection following successful DAA treatment over the three years of follow up. The study will also evaluate the proportion of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) with direct-acting anti-viral HCV therapy.

DETAILED DESCRIPTION:
In Australia, hepatitis C virus (HCV)-related morbidity and mortality have doubled in the past decade, with health care costs of $220 million per annum1. This is due to a large, ageing population with chronic infection (230,000), and low uptake of existing interferon-based therapy (1-2% per year) due to side-effects, and sub-optimal therapy efficacy. The majority of new (90%) and existing (80%) cases of HCV infection occur among people who inject drugs (PWID).

In the community, 15-20% of current PWID report recent (last month) receptive needle/syringe sharing2. Qualitative research shows that decisions about sharing equipment are multi-factorial and can include issues ranging from service access (such as distance to service and opening hours), concerns about anonymity, perceptions that HCV is ubiquitous and unavoidable3 to socially-located concerns that promote use of sterile equipment such as a desire to avoid "track marks"4. There is no research that examines sharing of injecting equipment in those with successful therapy in either community or prison settings.

Increasing access to HCV therapy is a key objective of national and NSW Hepatitis C Strategies5,6. The advent of well-tolerated, simple, oral hepatitis C virus (HCV) regimens - direct acting antivirals (DAAs) - has the potential to transform this landscape. These are much shorter, tolerable treatment regimens with cure >95%, providing an opportunity to reverse the rising burden of advanced liver disease. From 1st March 2016, these highly efficacious HCV therapies have been listed on the Pharmaceutical Benefit Scheme, and people with recent injecting drug use are eligible to receive them. This is an important feature of the listing. In many countries, people who have not ceased injecting drug use are ineligible to receive DAA therapy7, despite the fact that they comprise a significant proportion of HCV cases. Australia is therefore poised to lead the world in the scale-up of new therapies to an extent that many countries with such exclusions will not be able to achieve.

This feature of DAA access also affords unique opportunities with respect to the implementation of treatment scale-up in community drug treatment clinics. Australia has good treatment coverage for people who are opioid dependent, with over 50% of opioid dependent people estimated to engage in opioid substitution therapy (OST) 8. Community-based drug treatment clinics represent another logical venue for expansion of HCV care beyond existing tertiary HCV treatment centres 9,10.

Although response to DAA HCV therapy is high, lower responses have been observed among people with previous treatment experience9, cirrhosis9 and those with baseline or emergent resistance associated variants10. Such resistance associated variants can persist for up to two years after treatment11, affect re-treatment options12, and be transmitted to new hosts13. Further, PWID are likely to be exposed to multiple HCV infections as a result of ongoing high-risk behaviours and might commonly harbour mixed HCV infections (infection with two or more distinct viruses) 14. Underlying mixed HCV infection can contribute to nonresponse during therapy14, which has implications for DAA regimens that are preferentially active against specific viral genotypes or subtypes. These data argue for surveillance of HCV resistance and mixed HCV infection among PWID to resolve residual concerns regarding their clinical and public health significance.

Two systematic reviews assessing interferon-based therapy for PWID have demonstrated responses comparable to randomised controlled trials excluding PWID15, 16. These data have supported international recommendations for the management of HCV for PWID 17. However, there are limited data on DAA therapy among recent PWID. As treatment is broadened to include more marginalised individuals, many clinicians are reluctant to treat HCV among PWID with recent injecting drug use with new DAA therapies. Major concerns include poor adherence/response, increased risk behaviour and HCV reinfection.

A major concern is that ongoing injecting risk behaviours following DAA therapy in PWID will lead to HCV reinfection, reversing the benefits of cure. Ongoing risk behaviours following successful HCV therapy may lead to reinfection and compromised treatment outcomes14. In a systematic review and meta-analysis of HCV reinfection among PWID performed by the investigators, the pooled estimate of re-infection was 2.2/100 p-yrs (95% CI, 0.9-6.1) overall and 6.4/100 p-yrs (95% CI, 2.5-16.7) among individuals who reported injecting drug use post-SVR16. The one study of HCV reinfection post-therapy in prison performed to date was small (n=74), retrospective, and did not assess the rate of HCV reinfection18. Studies of reinfection following HCV therapy are limited by small sample sizes, retrospective study designs, incomplete follow-up, and a lack of sensitive methods to detect reinfection. Further, there are no data on HCV reinfection among recent PWID treated with DAAs.

Although DAA therapy could limit HCV-related disease burden, as treatment is broadened to include more marginalised individuals, many clinicians are reluctant to treat HCV among recent PWID, given concerns about poor adherence (and lower response to therapy), increased risk behaviours (due to the ease and high cure rates of DAA HCV therapy) and HCV reinfection (thereby reversing cure). However, no data exist on the extent to which this should be a concern. Given that DAA HCV therapy is highly expensive, we urgently need data on the magnitude of risk for, and predictors of, HCV reinfection. It is also unclear whether PWID treated in these two settings will vary in their response to DAA therapy and risk for reinfection.

The investigators have an excellent track record of conducting high quality cohort studies and clinical trials among PWID in the community19-23 and prison24, with high participant retention in follow-up. The investigators have developed a network of clinical sites providing HCV care in nine community-based drug treatment clinics20, 25. In SHARP-C the investigators will explore the risk of HCV reinfection and treatment efficacy among recent PWID with chronic HCV and recent injecting drug use.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have voluntarily signed the informed consent form.
2. Be ≥18 years of age on day of signing informed consent form.
3. Have chronic HCV infection.
4. Recent injecting drug use (previous 6 months).
5. Eligible for DAA therapy as per the Pharmaceutical Benefits Scheme (PBS) criteria
6. HIV-1 infected participants enrolled in the study must meet the following criteria:

   1. Have HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry (Baseline) and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load.
   2. Be on HIV Antiretroviral Therapy (ART) for at least 4 weeks prior to study entry using an ART regimen that is allowable with the intended DAA regimen as determined by the current PI and the Liverpool drug interaction website (http://www.hiv-druginteractions.org/) OR be naive to treatment with any antiretroviral therapy (ART) with a baseline CD4 count of >200 and have no plans to initiate ART treatment while participating in this study and through to at least Follow-up Week 4.

Exclusion Criteria:

1) The participant must be excluded from participating in the trial if the subject is unable or unwilling to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with chronic HCV infection and recent injecting drug use who are 18 years or over and are eligible for DAA therapy as per the PBS criteria.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Reinfection | 3 years
  Incidence of HCV reinfection following successful DAA therapy.

SECONDARY OUTCOMES:
Undetectable HCV RNA at SVR12 | 2.5 years
  The proportion of participants with a treatment response at SVR12
Treatment completion | 3 years
  The proportion of participants who complete treatment
Undetectable HCV RNA at the end of treatment | 3 years
  The proportion of participants with undetectable HCV RNA at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jason Grebely, Principal Investigator — Kirby Institute
Locations (4):
- Australia (4):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Drug and Alcohol Services (Hunter), Newcastle, New South Wales
  - Infectious Diseases Clinic, Royal Adelaide Hospital, Adelaide, South Australia